CLINICAL TRIAL: NCT03273439
Title: A Randomized, Double-blind Study of Repetitive Transcranial Magnetic Stimulation for Cognitive Deficits in Chronic Patients With Schizophrenia in a Chinese Han Population
Brief Title: A Study of rTMS for Cognitive Deficits in Chronic Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Psychiatric Hospital (Other)
Responsible Party: Principal Investigator, Zhe Li, Attending Psychiatrist, Suzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 46694276-1; Szzx201509 (Other Grant/Funding Number: Suzhou Key Medical Center for Psychiatric Diseases)
Record Dates: First submitted 2017-03-15; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia
Keywords: Repetitive transcranial magnetic stimulation; Negative symptoms; randomized controlled trial; Schizophrenia; cognition
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: In this study, we assessed the therapeutic effects and safety of left dorsolateral prefrontal cortex (DLPFC) high-frequency repetitive transcranial magnetic stimulation (rTMS) on negative symptoms of schizophrenia. We evaluated the efficacy of rTMS on cognition in patients with chronic schizophrenia.
Who Masked: Participant
Masking Description: This was a single-institution, randomized controlled, double blinded trial. Participants were randomized to receive, over 4 weeks, 20 sessions of either active or sham rTMS. Clinical assessment was performed at baseline, 4 weeks and 8 weeks by 2 psychiatrists blinded to the treatment assigned. Inter-rater reliability was satisfactory (κa=0.86).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- repetitive TMS (Experimental): Prior to each TMS administration, motor threshold was determined by stimulating the left motor strip with the lowest possible energy to produce, within 10 stimuli, at least 5 evoked potentials Z0.05 . In active rTMS, 10 Hz stimulations over left DLPFC occurred at a power of 110% of MT for 5-s intervals with 30-s intertrain interval. 30 trains were administered each day (MondayFriday) for 4 consecutive weeks (total stimuli=30,000).
  Interventions: Device: repetitive TMS
- Sham rTMS (Sham Comparator): all procedures were identical except they were the unmagnetized steel cylinders, instead of cylindrical magnets, that were rotated. Participants were, therefore, unable to distinguish between active and sham rTMS.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: repetitive TMS — Prior to each TMS administration, motor threshold was determined by stimulating the left motor strip with the lowest possible energy to produce, within 10 stimuli, at least 5 evoked potentials Z0.05 . In active rTMS, 10 Hz stimulations over left DLPFC occurred at a power of 110% of motor threshold (MT) for 5-s intervals with 30-s intertrain interval. 30 trains were administered each day (MondayFriday) for 4 consecutive weeks (total stimuli=30,000).
  Other Names: rTMS
  Arms: repetitive TMS
Device: Sham rTMS — Sham rTMS, without stimulation
  Arms: Sham rTMS

SUMMARY:
In this study, we assessed the therapeutic effects and safety of left dorsolateral prefrontal cortex (DLPFC) high-frequency repetitive transcranial magnetic stimulation (rTMS) on negative symptoms of schizophrenia. We evaluated the efficacy of rTMS on cognition in patients with chronic schizophrenia.

DETAILED DESCRIPTION:
This is a randomized, sham-controlled, double-blinded trial. 47 patients diagnosed with schizophrenia on stable antipsychotic treatment were randomly assigned to active rTMS treatment group (n=25) or a sham rTMS treatment group (n=22). 25 patients in the active rTMS group received 10 Hz 110% rTMS, while 22 patients were subjected to sham rTMS, both being given 4-week treatment (5 days per week). Efficacy of negative symptom was assessed with the Scale for the Assessment of Negative Symptoms (SANS), the Positive and Negative symptom scale (PANSS) at baseline, the end of 4 weeks and 8 weeks. The cognitive function was assessed with CANTAB at baseline, the end of 4 weeks and 8 weeks .The side effects were assessed with Treatment Emergent Symptoms Scale at baseline and the end of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Right-handed;
2. meeting the diagnosis of schizophrenia for at least 2 years;
3. had been on anti-psychotic medications for more than 12 weeks;
4. with unresolved negative symptoms (SANS>20).

Exclusion Criteria:

1. with substance use disorders ;
2. with cerebral pathologies (e.g. seizure, aneurysm, stroke), intra-cranial metals, pacemakers, severe cardiovascular diseases;
3. receiving electroconvulsive therapy in the past 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Scale for the Assessment of Negative Symptoms (SANS) | 4 weeks
  clinical negative symptoms

SECONDARY OUTCOMES:
Positive and Negative symptom scale (PANSS) | 4 weeks
  Clinical symptoms
CANTAB | 4 weeks
  cognition

CONTACTS AND LOCATIONS:
Overall Officials: Guangzhong Yin, MD, Study Chair — Suzhou Guangji Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Lu X, Du S, Hu W, Xiao D, He B, Su C, Lin S, Zhan Q, Wu H, Li Z. Effects of varied rTMS frequencies on cognitive function in individuals with chronic schizophrenia: A double-blind randomized controlled trial. J Psychiatr Res. 2025 Sep;189:33-41. doi: 10.1016/j.jpsychires.2025.05.052. Epub 2025 May 23. PMID 40479952